CLINICAL TRIAL: NCT05130125
Title: Retrospective Cohort Observational Study to Evaluate the Effectiveness and Safety of Fresh or Frozen Embryo Transfer After Ovarian Hyperstimulation (Administration of rFSH or HP-hMG Alone or Co-administration of rFSH and HP-hMG)
Brief Title: Retrospective Cohort Observational Study to Evaluate the Effectiveness and Safety of Fresh or Frozen Embryo Transfer
Status: Completed | Type: Observational
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Other Study IDs: LG-IMHOS001
Record Dates: First submitted 2021-11-04; First posted 2021-11-22 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2021-11

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fresh embryo: fresh embryo transfer after ovarian hyperstimulation
  Interventions: Drug: rFSH
- frozen embryo: frozen embryo transfer after ovarian hyperstimulation
  Interventions: Drug: rFSH

INTERVENTIONS:
Drug: rFSH — rFSH or HP-hMG or rFSH and HP-hMG
  Other Names: HP-hMG; rFSH and HP-hMG

SUMMARY:
A multicenter, retrospective cohort observational study to evaluate the effectiveness and safety of fresh or frozen embryo transfer after ovarian hyperstimulation (administration of rFSH or HP-hMG alone or co-administration of rFSH and HP-hMG)

DETAILED DESCRIPTION:
A multicenter, retrospective cohort observational study to evaluate the effectiveness and safety of fresh or frozen embryo transfer after ovarian hyperstimulation (administration of rFSH or HP-hMG alone or co-administration of rFSH and HP-hMG) to infertile female patients undergoing assisted reproductive technology to controlled ovarian hyperstimulation

ELIGIBILITY:
Inclusion Criteria:

* First IVF-ET cycle patients

Exclusion Criteria:

Poor ovarian responder

- At least two of the following three features must be present: (i) Advanced maternal age (≥ 40 years) or any other risk factor for Poor ovarian response (POR); (ii) A previous POR (≤ 3 oocytes with a conventional stimulation protocol); (iii) An abnormal ovarian reserve test (i.e. AFC < 5-7 follicles or AMH < 0.5-1.1 ng/mL)

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: infertile female patients
Sampling Method: Probability Sample
Enrollment: 1166 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Oocytes | average of 14 days
  Counting number of Oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Jieun Shin, Principal Investigator — Cha medical center
Locations (1):
- CHA Fertility Hospital, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No